CLINICAL TRIAL: NCT01911923
Title: Reduction in Postoperative Atelectasis by Continuous Positive Airway Pressure and Low Oxygen Concentration After Endotracheal Extubation.
Brief Title: Ventilation Strategy Reduces Postoperative Atelectasis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Region Västmanland (Other)
Responsible Party: Principal Investigator, Lennart Edmark, M.D., Region Västmanland
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dnr 2008 / 251
Record Dates: First submitted 2013-07-26; First posted 2013-07-30 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2014-08

CONDITIONS: Pulmonary Atelectasis
MeSH Terms: conditions — Pulmonary Atelectasis | interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No CPAP/PEEP and 100 % oxygen (Active Comparator): This is the control group
  Interventions: Procedure: No CPAP/PEEP and 100 % oxygen
- CPAP/PEEP and 30 % oxygen (Experimental): This is the intervention group
  Interventions: Procedure: CPAP/PEEP and 30 % oxygen

INTERVENTIONS:
Procedure: No CPAP/PEEP and 100 % oxygen — This is the control group and 100 % oxygen will be used during induction of and emergence from anesthesia, no enhanced level of CPAP/PEEP is implemented. During controlled ventilation ventilation mode is volume controlled.
  Arms: No CPAP/PEEP and 100 % oxygen
Procedure: CPAP/PEEP and 30 % oxygen — During all phases of anesthesia CPAP/PEEP will be used together with 100 % oxygen during induction of as well during emergence from anesthesia until after extubation when 30 % oxygen will be used.
  Arms: CPAP/PEEP and 30 % oxygen

SUMMARY:
Atelectasis is common during and after general anesthesia. The investigators hypothesized that a ventilation strategy with a combination of 1) continuous positive airway pressure (CPAP) or positive end-expiratory pressure (PEEP) and 2) a reduced end-expiratory oxygen fraction (FETO2) before commencing mask ventilation with CPAP after extubation would reduce the area of postoperative atelectasis.

DETAILED DESCRIPTION:
During general anesthesia, the combination of reduced functional residual capacity (FRC), high inspiratory oxygen fraction (FIO2), and airway closure are the main factors implicated in the atelectasis, shunt and shunt-like effects that account for the majority of the impaired oxygenation seen during general anesthesia.

Previous studies have shown that formation of atelectasis during preoxygenation and induction of anesthesia can be avoided by adding a continuous positive airway pressure (CPAP) followed by a positive end-expiratory pressure (PEEP).During emergence from anesthesia, high concentrations of oxygen predispose to atelectasis formation. Even a recruitment maneuver, followed by ventilation with 100% oxygen with a PEEP/CPAP of 10 cm H2O until extubation, failed to improve postoperative oxygenation compared with that achieved with zero end-expiratory pressure (ZEEP).This failure may have been caused by the presence of lung regions with high oxygen concentrations.

The investigators hypothesized that by inducing and discontinuing anesthesia during CPAP/PEEP and deliberately reducing FIO2 after extubation, postoperative atelectasis would be reduced compared with standard protocols. To test our hypothesis, the investigators studied 1) a control group with no CPAP/PEEP and a FIO2 of 1.0 while breathing spontaneously after extubation, and 2) an intervention group that was on CPAP/PEEP of 6 cmH2O from induction to extubation and that received an FIO2 of 1.0 until extubation and then an FIO2 of 0.3 via a facemask while on CPAP after extubation.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients up to 75 years of age.
2. American Society of Anesthesiologists (ASA) physical status class I-III.
3. Be able to climb two flight of stairs without stopping.
4. SpO2 of ≥ 94% when breathing air in the supine position.
5. A body mass index (BMI, weight in kilograms divided by the square of the height in meters) of < 31.

Exclusion Criteria:

1. Patients with chronic obstructive pulmonary disease.
2. Smokers.
3. Ex smokers if smoked more than 5 pack years.
4. Overt heart failure
5. Known or predicted difficult intubation.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-08; Primary Completion 2013-11 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Area of atelectasis | 30 minutes
  The area of atelectasis is investigated by computed tomography of the lungs postoperatively

SECONDARY OUTCOMES:
Peripheral oxygen saturation (SpO2) | 2 hours
  SpO2 is assessed immediately after extubation and then continuously postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Lennart Edmark, Md, Principal Investigator — Landstinget Vastmaland
Locations (1):
- Västmanlands sjukhus Köping, Köping, Västmanland County, Sweden